CLINICAL TRIAL: NCT01386840
Title: IndiaCLEN Multicentric Trial of Home Versus Hospital Oral Amoxicillin for Management of Severe Pneumonia in Children
Brief Title: IndiaCLEN Multicentre Trial of Home Versus Hospital Oral Amoxicillin for Management of Severe Pneumonia in Children
Acronym: ISPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lata Medical Research Foundation, Nagpur (Other)
Collaborators: Indira Gandhi Medical College, Shimla (Other); International Clinical Epidemiology Network (INCLEN) TRUST (Network); MCH-STAR Initiative, India (Unknown)
Responsible Party: Principal Investigator, Dr.Archana B Patel, Professor, Pediatrics, Lata Medical Research Foundation, Nagpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02_ISPOT
Record Dates: First submitted 2011-06-25; First posted 2011-07-01 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Pneumonia
Keywords: Efficacy of Treatment; Severe; home treatment; treatment at hospital
MeSH Terms: conditions — Pneumonia; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Severe Pneumonia - Hospital Management (No Intervention): Those randomized to hospital management will be monitored by health personnel for at least 48 hours for clinical deterioration and parameters like temperature, Respiratory rate, Lower chest indrawing, Pulse rate, Clinical deterioration, Other signs eg. comorbid conditions, Assessment of adherence, Adverse event.
  Mothers, whose children are discharged after 48 hours, will be counseled to continue with oral treatment prescribed for a period of 7 days and will be advised to return to healthcare facility at their scheduled times and any time during the study period if there is clinical deterioration. The symptoms and signs of clinical deterioration will be discussed with the mother as described in the "patient discharge counselling checklist". Mothers will be given a "study patient data card"
- Severe Pneumonia - Home Management (Experimental): For those randomized to home management, first dose will be administered by the mother/caretaker under supervision at health facility. The health personnel will assess the parameters like temperature, Respiratory rate, Lower chest indrawing, Pulse rate, clinical deterioration, Other signs eg. co-morbid conditions, Assessment of adherence, Adverse event when they visit the home after 24 hours, 72 hours and on day 8th.
  Mothers will be advised to return to the healthcare facility at their scheduled times and any time during the study period if there is clinical deterioration. The symptoms and signs of clinical deterioration will be discussed with the mother as described in the "patient discharge counselling checklist". Mothers will be given a "study patient data card" with contact Numbers.
  Interventions: Other: Severe Pneumonia - Home Management

INTERVENTIONS:
Other: Severe Pneumonia - Home Management — For those randomized to home management, first dose will be administered by the mother/caretaker under supervision at health facility. The health personnel will assess the parameters like temperature, Respiratory rate, Lower chest indrawing, Pulse rate, clinical deterioration, Other signs eg. co-morbid conditions, Assessment of adherence, Adverse event when they visit the home after 24 hours, 72 hours and on day 8th.
  Mothers will be advised to return to the healthcare facility at their scheduled times and any time during the study period if there is clinical deterioration. The symptoms and signs of clinical deterioration will be discussed with the mother as described in the "patient discharge counselling checklist". Mothers will be given a "study patient data card" with contact Numbers.
  Arms: Severe Pneumonia - Home Management

SUMMARY:
The purpose of this study is to determine the safety and efficacy of oral amoxicillin in treating WHO defined severe pneumonia(cough and fast breathing with lower chest indrawing) at home and at hospital using an open labelled multicentric prospective two-arm randomized clinical trial to determine the differences in failure of treatment with a 7 day course of oral amoxicillin administered for first 48 hours in the hospital in comparison to being sent home after enrolment, in children 3 to 59 months old who have severe pneumonia. The investigators developmental hypothesis were to test whether the community/home based oral amoxicillin is efficacious for treating severe pneumonia.

DETAILED DESCRIPTION:
Primary objectives of this trial are to assess the rates of treatment failure (as defined below) within the first 7 days or efficacy of a 7 day course of oral amoxycillin when administered at home in comparison to administration of oral amoxycillin for first 48 hours in the hospital.

Treatment failure is defined as follows-

* Clinical deterioration of disease any time after enrollment: developing any sign of very severe disease such as persistent vomiting (vomiting repeated thrice within an hour due to any reason), central cyanosis, grunt, stridor, abnormally sleepy or difficult to wake, inability to drink, convulsions, or death.
* Change of antibiotic: due to persistent vomiting (vomiting of amoxycillin within 20 minutes of administration; 3 such attempts), or, developing a co-morbid condition, or persisting fever > 98.6°F with lower chest indrawing even after 3rd day, or, fever alone at or after day 5, or, lower chest indrawing alone (non responsive to three doses of nebulization with bronchodilator) at or after day 5(as reported by the mother), or, persistence of fast breathing after day 7 which is non responsive to three doses of nebulisation with bronchodilator.
* Hospitalization: any time in home managed patients or clinical decision to extend the hospitalization longer than 48 hours in hospitalized children or re-hospitalization in those discharged after 48 hours from hospital. It could be related to pneumonia, or to therapy with amoxycillin [relatedness determined by the Data & Safety Monitoring Board (DSMB)].
* Children who need to restart antibiotics i.e. "failure of treatment", between day 8th and day 14th due to reappearance of any danger signs, lower chest indrawing or fast breathing which is non responsive to three trials of nebulization with bronchodilator.
* Serious adverse event considered possibly or probably related to amoxycillin.
* Left against medical advice (LAMA) or Voluntary withdrawal of consent from study from enrollment uptill day 14th.
* Loss to follow up uptill day 14th.

Secondary objectives of this trial are to determine in children receiving oral amoxycillin for severe pneumonia, the following:

* Determine the proportion of children who need to restart antibiotics i.e. "failure of treatment", between day 8th and day 14th due to reappearance of any danger signs, lower chest indrawing or fast breathing which is non responsive to three trials of nebulization with bronchodilator.
* To identify clinical predictors at baseline and during the course of treatment that predicts "failure of oral treatment", from enrollment till day 14th.
* The costs of home and hospital management of severe pneumonia with oral amoxycillin.
* Left against medical advice (LAMA) or Voluntary withdrawal of consent from day 7th to day 14th.
* Loss to follow up from day 8th to day 14th.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 59 months with pneumonia and lower chest wall indrawing
* Ability to take orally
* Absence of radiological consolidation or effusion
* Informed consent by a legal guardian

Exclusion Criteria:

Children with any of the following conditions:

* Very severe pneumonia/disease
* Respiratory rate > 70/min
* Persistent vomiting
* Known prior episodes of asthma, or, three or more prior episodes of wheezing
* LCI that resolves after three doses of bronchodilator therapy1
* Documented use of prior oral antibiotics for 48 hours
* Severe malnutrition (weight for height < 3SD or kwashiorkor)
* Known penicillin or amoxicillin allergy
* Hospitalization in the last two weeks
* Known or clinically recognizable HIV, congenital cardiac or respiratory anomalies, chronic lung disease including bronchopulmonary dysplasia, neurological impairment that affects respiratory function, renal diseases, malignant or haematological diseases.
* Other diseases requiring antibiotic therapy at presentation, such as meningitis,dysentery, osteomyelitis, septic arthritis, evident tuberculosis, etc.
* Anaemia requiring blood transfusion
* Kerosene poisoning
* Measles in the last 15 days
* Previous inclusion in the study or already included in another study
* Living outside a pre-defined area
* Parental or caretaker refusal to participate in the study

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1118 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of a 7 day course of oral amoxycillin when administered at Home in comparison to administration of oral amoxycillin for first 48 hours in the hospital | Day of enrollment to Day 7
  Primary outcomes are to assess the efficacy of a 7 day course of oral amoxycillin when administered at home in comparison to administration of oral amoxycillin for first 48 hours in the hospital, on the following study outcomes, the presence of any one of which indicate "failure of treatment" :
  * Clinical deterioration of disease any time after enrollment
  * Change of antibiotic
  * Hospitalization
  * Serious adverse event considered possibly or probably related to amoxycillin.
  * Left against medical advice (LAMA)
  * Loss to follow up on day 8th

SECONDARY OUTCOMES:
To determine factors leading to treatment failure from day 8 to day 14 and costs of home and hospital management of severe pneumonia with oral amoxycillin | Day 8 to Day 14
  Secondary outcome of this trial are to determine the following:
  * Determine the proportion of children who need to restart antibiotics i.e. "failure of treatment", between day 8th and day 14th due to reappearance of any danger signs, lower chest indrawing or fast breathing
  * To identify clinical predictors at baseline and during the course of treatment that predicts "failure of oral treatment",
  * The costs of home and hospital management of severe pneumonia with oral amoxycillin.
  * Left against medical advice (LAMA)
  * Loss to follow up from day 8th to day 14th.

CONTACTS AND LOCATIONS:
Overall Officials: Archana B Patel, MD,DNB,PhD, Principal Investigator — Professor And Head, Pediatrics, Indira Gandhi Govt. Medical College & CEO and Vice President, Lata MEdical Research Foundation, Nagpur
Locations (6):
- India (6):
  - Post Graduate Institute of Medical Sciences, Chandigarh, Chandigarh, Chandigarh
  - Indira Gandhi Govt. Medical College, Nagpur, Nagpur, Maharashtra
  - B.J. Medical College, Pune, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sevagram, Wardha, Maharashtra
  - Institute of Child Health, Chennai, Chennai, Tamil Nadu
  - Jawaharlal Nehru Medical College, Aligarh Muslim University, Aligarh, Uttar Pradesh

REFERENCES:
- [Derived] Patel AB, Bang A, Singh M, Dhande L, Chelliah LR, Malik A, Khadse S; ISPOT Study Group. A randomized controlled trial of hospital versus home based therapy with oral amoxicillin for severe pneumonia in children aged 3 - 59 months: The IndiaCLEN Severe Pneumonia Oral Therapy (ISPOT) Study. BMC Pediatr. 2015 Nov 17;15:186. doi: 10.1186/s12887-015-0510-9. PMID 26577943